CLINICAL TRIAL: NCT00989820
Title: Efficacy of Adding Hyperbaric Oxygen Therapy to the Treatment of Late Radiation Damage of the Lower Jaw (Osteoradionecrosis).
Brief Title: Efficacy of Hyperbaric Oxygen Therapy in the Treatment of Osteoradionecrosis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment problems, patients refused to participate
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL20963.091.08
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2020-12

CONDITIONS: Osteoradionecrosis
Keywords: osteoradionecrosis; mandible; radiotherapy; hyperbaric oxygen therapy
MeSH Terms: conditions — Osteoradionecrosis | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (No Intervention): This is the standard arm. Surgery without hyperbaric oxygen treatment
- Hyperbaric oxygen therapy with surgery (Experimental): Intervention arm. Hyperbaric oxygen therapy with surgery.
  Interventions: Drug: hyperbaric oxygen

INTERVENTIONS:
Drug: hyperbaric oxygen — 30 session inhalation of 100% oxygen in a pressure chamber under 2.4 ATA for 90 minutes a day before surgery and 10 session hyperbaric oxygen therapy (as mentioned before) after surgery
  Other Names: Linde Gas Therapeutics Benelux B.V.; RVG 30355; ATC code V03AN012
  Arms: Hyperbaric oxygen therapy with surgery

SUMMARY:
The purpose of this study is to determine whether hyperbaric oxygen therapy is effective in the treatment of osteoradionecrosis (late complication of radiation therapy) of the jaw.

DETAILED DESCRIPTION:
Damage to the lower jaw as a late complication of radiation therapy (osteoradionecrosis (ORN)) is often seen in patients treated with radiation therapy for a tumor in the head and neck region. Part of the lower jaw becomes non-vital and has to be treated. ORN proofs to be a condition difficult to treat and the treatment for this condition varies.

In many countries hyperbaric oxygen therapy (HBOT) is added to the surgical treatment of ORN. Unfortunately there is no consensus whether the addition of hyperbaric oxygen therapy to the treatment of ORN is beneficial or not. This study has the aim to investigate the efficacy and cost-effectiveness of HBOT in the treatment of ORN.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age ≥ 18 jr
* WHO performance status 0-2
* Last radiation treatment ≥ 6 month ago radiotherapy with curative intention and > 55 Gy. The affected part of the jaw must be in the target volume area of the radiotherapy field.
* Local recurrence must be ruled out
* Necrosis of the jaw with at least one of the following symptoms for over 3 month present:

  * Bone exposition which measures at least 1 cm
  * Evident bone lesions at radiologic evaluation (panorex) that fits the diagnosis ORN.
  * Non-healing extraction socket

Exclusion Criteria:

* Former HBO treatment
* Contra indication for HBO treatment (pneumothorax)
* Bisphosphonate treatment in the medical history
* reirradiation in the medical history
* Osteosynthesis material in the affected area
* Distant metastasis
* Primary or recurrent tumor in the affected area
* Malignancies elsewhere

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
absence of exposed bone, fistulae or ulceration. | 12 months after finishing therapy in the arm assigned to
  Number of patients with complete healing

SECONDARY OUTCOMES:
Pain score | one year after therapy in the arm assigned to.
  VAS 0-10 (0 absence of pain, 10 unbearable pain)
Clinical and radiological assessment of the treatment response | one year after therapy in the arm assigned to.
  Light photography and X-rays to assess the amount of patients without mucosal or bone lesions one year after therapy. The measurements between the start and finish of the inclusion are used to assess increase or decline of the lesions during therapy
Completion of the therapy in the arm for which patient has been randomized; if someone drops out of this study the reason will be scored. | one year after therapy in the arm assigned to.
  Drop out rate of included patients and scoring of the reason for termination before completing the study.
Use of pain medication | one year after therapy in the arm assigned to.
  type and quantity
Type of surgical intervention | one year after therapy in the arm assigned to.
  For each individual patient the type of surgery is scored: sequestrectomy, marginal mandibula resection, segment resection
Quality of life | one year after therapy in the arm assigned to.
  Quality of life questionnaires EORTC-QoL-C30, Head and Neck-C35. These QoL questionaires are for general QoL for oncology patients (C-30) with a specific part for head and neck oncology (C-35)
Cost effectiveness | one year after therapy in the arm assigned to.
  Questionnaire EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Francois Dieleman, MD DMD, Principal Investigator — Radboud University Medical Center; Thijs Merkx, MD DMD PhD, Study Director — Radboud University Medical Center; Hans Kaanders, MD PhD, Study Director — Raboud University Medical Centre
Locations (8):
- Netherlands (8):
  - NKI/AvL, Amsterdam
  - VU University Medical centre, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht Universitary Medical Centre, Maastricht
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Erasmus University Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- See also: Dutch Co-operative Head and Neck Group — http://www.nwhht.nl